CLINICAL TRIAL: NCT01367964
Title: Early Treatment of Infants at High Risk of Developing West Syndrome With Low-dose Adrenocorticotropin Hormone (ACTH)
Brief Title: Prevention of West Syndrome With Low-dose Adrenocorticotropin Hormone (ACTH)
Acronym: PREVENT-WS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, John J Millichap, MD, Attending Physician, Division of Neurology, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2011-14518
Record Dates: First submitted 2011-06-03; First posted 2011-06-07 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: West Syndrome
Keywords: Hypsarrhythmia; Spasms, Infantile; West Syndrome
MeSH Terms: conditions — Spasms, Infantile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACTH treatment (Experimental): Infants with a Type 3 EEG (pre-hypsarhythmia) will be treated with ACTH for 2 weeks.
  Interventions: Drug: adrenocorticotropin hormone

INTERVENTIONS:
Drug: adrenocorticotropin hormone — ACTH 16 units intramuscular injection once daily for 2 weeks
  Other Names: H.P. Acthar® Gel (repository corticotropin injection)

SUMMARY:
West syndrome (WS) is a specific type of epilepsy (or seizure disorder) that has three features: infantile spasms (type of seizure), loss of milestones, and a specific pattern on electroencephalogram (EEG or brain wave test) called hypsarhythmia. The purpose of this study is to detect pre-hypsarhythmia in infants at high-risk for WS and determine whether treatment with ACTH will prevent WS.

DETAILED DESCRIPTION:
Hypothesis: Preemptive ACTH will halt the evolution of hypsarhythmia and improve the EEG patterns in infants with pre-hypsarhythmic EEG.

Aim. To determine whether a low dose ACTH improves EEG, we will repeat EEG one month after a 2 week course of daily ACTH.

ELIGIBILITY:
Inclusion criteria:

* Infants with pre-hypsarhythmia (Type 3 EEG) between 2 months to 12 months of age.

Exclusion criteria:

* Infants with any of the following diagnoses:
* A previous history of infantile spasms;
* Known inborn error of metabolism;
* Other symptomatic epileptic encephalopathy (e.g. Ohtahara syndrome).

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2011-07; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Evidence for improvement in the EEG one month following initiation of the 2 week course of low-dose ACTH. | 1 month
  If pre-hypsarhythmia (Type 3) is detected, ACTH treatment is given for 2 weeks and an EEG is performed one month later. Primary outcome is improvement in EEG (as defined by assigned type).

CONTACTS AND LOCATIONS:
Overall Officials: John J. Millichap, MD, Principal Investigator — Ann & Robert H. Lurie Children's Hospital of Chicago and Northwestern University Feinberg School of Medicine; Sookyong Koh, MD, PhD, Principal Investigator — Ann & Robert H. Lurie Children's Hospital of Chicago and Northwestern University Feinberg School of Medicine; Doulgas R Nordli, Jr, MD, Principal Investigator — Ann & Robert H. Lurie Children's Hospital of Chicago and Northwestern University Feinberg School of Medicine
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] SOREL L, DUSAUCY-BAULOYE A. [Findings in 21 cases of Gibbs' hypsarrhythmia; spectacular effectiveness of ACTH]. Acta Neurol Psychiatr Belg. 1958 Feb;58(2):130-41. No abstract available. French. PMID 13532578
- [Background] Okumura A, Watanabe K. Clinico-electrical evolution in pre-hypsarrhythmic stage: towards prediction and prevention of West syndrome. Brain Dev. 2001 Nov;23(7):482-7. doi: 10.1016/s0387-7604(01)00291-1. PMID 11701242
- [Background] Suzuki M, Okumura A, Watanabe K, Negoro T, Hayakawa F, Kato T, Itomi K, Kubota T, Maruyama K. The predictive value of electroencephalogram during early infancy for later development of West syndrome in infants with cystic periventricular leukomalacia. Epilepsia. 2003 Mar;44(3):443-6. doi: 10.1046/j.1528-1157.2003.29202.x. PMID 12614401
- [Background] Philippi H, Wohlrab G, Bettendorf U, Borusiak P, Kluger G, Strobl K, Bast T. Electroencephalographic evolution of hypsarrhythmia: toward an early treatment option. Epilepsia. 2008 Nov;49(11):1859-64. doi: 10.1111/j.1528-1167.2008.01715.x. Epub 2008 Jul 9. PMID 18631366
- [Background] Watanabe K, Iwase K, Hara K. The evolution of EEG features in infantile spasms: a prospective study. Dev Med Child Neurol. 1973 Oct;15(5):584-96. doi: 10.1111/j.1469-8749.1973.tb05169.x. No abstract available. PMID 4358106
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- See also: Lurie Children's Epilepsy Center — https://www.luriechildrens.org/en/specialties-conditions/pediatric-epilepsy/